CLINICAL TRIAL: NCT04618809
Title: Improving the Approach to and Management of the Older Patient With Metastatic Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Efrat Dotan, Efrat Dotan, MD, Fox Chase Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-8006
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Provider Didactic Intervention (Experimental): * Phase 1 - Providers complete a needs assessment questionnaire, which evaluates the approach to older mGC patients at each site.
  * Phase 2 - Providers participate in an hour-long didactic session and begin enrolling eligible metastatic gastric cancer (mGC) patients. Enrolled mGC patients complete a comprehensive geriatric assessment (CGA). Providers complete the treatment plan and review of geriatric assessment questionnaires, which also includes an evaluation of their overall view of the utility of the geriatric assessment.
  * Phase 3 - Follow-up chart reviews (2-3 months post intervention) are completed to assess for actual implementation of recommended interventions identified by the geriatric assessment.
  Interventions: Behavioral: Didactic Session; Behavioral: Comprehensive Geriatric Assessment, including an exploratory analysis to evaluate the use of fitness trackers for evaluation of functional status.

INTERVENTIONS:
Behavioral: Didactic Session — This session will include an overview of the approach to and management of older mGC patients patients through a case-based presentation.
Behavioral: Comprehensive Geriatric Assessment, including an exploratory analysis to evaluate the use of fitness trackers for evaluation of functional status. — * The Comprehensive Geriatric Assessment (CGA) is a composite of assessment scales evaluating physical, psychological, and social well-being, and is the recommended tool for evaluating an older cancer patient and determining appropriateness of therapy.
  * The patient will receive a FitBit TM to wear for 4 days. Number of steps/day will be recorded.

SUMMARY:
The purpose of this study is to enhance the care of older metastatic gastric cancer (mGC) patients by increasing awareness among oncology providers of the unique aspects of care required for older patients. The goal of the study is to educate providers on the utility of geriatric assessment in guiding therapy of older mGC patients. The investigators will also assess the feasibility and benefit of incorporating geriatric self-assessments into clinical practice. The study will include four phases.

DETAILED DESCRIPTION:
Older oncology patients pose a significant treatment challenge due to poor chemotherapy tolerance as a result of underlying co-morbidities, lack of social support, and diminished functional reserve. Oncologists are faced with the challenge of differentiating between patients that can and cannot tolerate chemotherapy, and tailoring therapy to the patient's biologic rather than chronologic age.

A significant challenge that surrounds the treatment of the older metastatic gastric cancer (mGC) patient in particular, lies in the lack of evidence based clinical data to guide the oncologist in determination of a treatment plan. This is a result of under representation of older patients in clinical trials. Due to these challenges, a thorough evaluation of the older patient is recommended prior to initiation of anti-cancer therapy.

The purpose of this research study is to enhance the care of the older mGC patient by increasing awareness among oncology providers of the unique aspects of care required for older patients. The goal of the study is to educate providers on the utility of geriatric assessment in guiding therapy of older metastatic gastric cancer patients. The investigators will also assess the feasibility and benefit of incorporating geriatric self-assessments into clinical practice. The study will include four phases:

1. Needs assessments - to understand the population of older gastric cancer patients seen in routine practice at community and academic centers, and assess their treatment approach.
2. Educational programming about management of older metastatic gastric cancer patients, and geriatric assessment of these patients.
3. Active testing of the use of geriatric assessment in clinical practice, including an exploratory analysis to evaluate the use of fitness trackers for evaluation of functional status.
4. Short-term follow-up chart reviews (2-3 months post intervention) to assess for actual implementation of recommended interventions identified by the geriatric assessment.

The ultimate goal is to expand this educational intervention to other oncology practices beyond those participating in this study, and for all older cancer patients regardless of their disease site. During this study period we will identify the specific gaps that exist in each practice for the care of older patients with mGC. This information is crucial to understand the needs of this patient population and will inform future trials with possible intervention. The second phase of our study will expose the practices to the use of a geriatric assessment through a patient's self-assessment tool and demonstrate its feasibility. Our hope is that all involved practices will find benefit from incorporating a geriatric assessment into their practice and will continue to use it in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to read and understand English, ability to sign consent, and complete a self-assessment evaluation.
2. Evidence of mGC (mGE junction cancer allowed). Patients can be enrolled at any stage of their treatment or disease course.
3. Ongoing active therapy for mGC. Patients can be treated with any type of therapy including chemotherapy, immunotherapy or Her-2 targeted therapy.
4. Life expectancy ≥3 months.

Exclusion Criteria:

1. ≤69 years old.
2. Inability to read and understand English.
3. No evidence of mGC.
4. Not on active therapy.
5. Life expectancy <3 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of geriatric abnormalities detected. (Tool used: Comprehensive Geriatric Assessment) | 18 Months
  Investigators will test the proportions of patients having at least one abnormality detected by the Comprehensive Geriatric Assessment that was missed in the standard clinical assessment compared to a null-hypothesis rate of 5%.
  The Comprehensive Geriatric Assessment includes the following scales:
  Eastern Cooperative Oncology Group Performance Status, Self-rated Performance Status, Katz Activities of Daily Living scale, Lawton Instrumental Activities of Daily Live Scale, Timed Up and Go, Number of Falls in past 6 months, Medical Social Support Scale, Geriatric Depression Scale, National Comprehensive Cancer Center Distress Thermometer, Blessed Orientation Memory Concentration Scale, Charlson Comorbidity Index, Body Mass index,Mini Nutritional Assessment, Cancer and Aging Research Group Chemotherapy Toxicity Prediction Calculator, Comprehensive Score for Financial Toxicity - Functional Assessment of Chronic Illness Therapy scale
Percentage of treatment plan changes. (Count # of treatment changes 2-3 months after comprehensive geriatric assessment. Site coordinators will complete follow-up chart review of each patient to see what, if any, changes were made) | 18 months
  Investigators will assess the percentage of physician reported cases whose treatment plan was modified due to responses on the Comprehensive Geriatric Assessment.

SECONDARY OUTCOMES:
Provider perception (Review of Geriatric Assessment Questionnaire) | 18 months
  Measurement of provider perception of the efficacy and feasibility of the didactic educational session via questionnaire
Fitbit assessed functional status. Fitbit data: step count | 18 months
  We aim to determine the feasibility of using fitbits in this patient population and evaluate the correlation between step count, physician recorded performance status, and scores on functional assessment in the comprehensive geriatric assessment.
  We will compare data collected from the FitBit to both the physician-reported and CGA-identified functional status (Timed Up and Go, Activities of Daily Living, Instrumental Activities of Daily Living, and number of falls in the past 6 months) in each patient.
Fitbit assessed functional status. Fitbit data: distance logged | 18 months
  We aim to determine the feasibility of using fitbits in this patient population and evaluate the correlation between distance logged, physician recorded performance status, and scores on functional assessment in the comprehensive geriatric assessment.
  We will compare data collected from the FitBit to both the physician-reported and CGA-identified functional status (Timed Up and Go, Activities of Daily Living, Instrumental Activities of Daily Living, and number of falls in the past 6 months) in each patient.
Fitbit assessed functional status. Fitbit data: moderately active, lightly active, and sedentary minute categorization. | 18 months
  We aim to determine the feasibility of using fitbits in this patient population and evaluate the correlation between moderately active, lightly active, and sedentary minute categorization, physician recorded performance status, and scores on functional assessment in the comprehensive geriatric assessment.
  We will compare data collected from the FitBit to both the physician-reported and CGA-identified functional status (Timed Up and Go, Activities of Daily Living, Instrumental Activities of Daily Living, and number of falls in the past 6 months) in each patient.
Fitbit assessed functional status. Fitbit data: floors climbed | 18 months
  We aim to determine the feasibility of using fitbits in this patient population and evaluate the correlation between floors climbed, physician recorded performance status, and scores on functional assessment in the comprehensive geriatric assessment.
  We will compare data collected from the FitBit to both the physician-reported and CGA-identified functional status (Timed Up and Go, Activities of Daily Living, Instrumental Activities of Daily Living, and number of falls in the past 6 months) in each patient.
Fitbit assessed functional status. Fitbit data: calories burned | 18 months
  We aim to determine the feasibility of using fitbits in this patient population and evaluate the correlation between calories burned, physician recorded performance status, and scores on functional assessment in the comprehensive geriatric assessment.
  We will compare data collected from the FitBit to both the physician-reported and CGA-identified functional status (Timed Up and Go, Activities of Daily Living, Instrumental Activities of Daily Living, and number of falls in the past 6 months) in each patient.
Fitbit assessed functional status. Fitbit data: heart rate | 18 months
  We aim to determine the feasibility of using fitbits in this patient population and evaluate the correlation between heart rate, physician recorded performance status, and scores on functional assessment in the comprehensive geriatric assessment.
  We will compare data collected from the FitBit to both the physician-reported and CGA-identified functional status (Timed Up and Go, Activities of Daily Living, Instrumental Activities of Daily Living, and number of falls in the past 6 months) in each patient.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania